CLINICAL TRIAL: NCT06219850
Title: Effectiveness of a Physical Exercise and Nutritional Education Strategy on Physical Fitness and Cardiometabolic Health in People With Type 2 Diabetes Mellitus: Longitudinal Design of the EDUGUTION Study
Brief Title: Physical Exercise, Diet, and Health in People With Type 2 Diabetes: Longitudinal Design of the EDUGUTION Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cadiz (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Other Study IDs: EDUGUTION YEAR
Record Dates: First submitted 2023-10-03; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Fat Burn; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Metabolism Disorder
Keywords: exercise; diet; metabolism; physical fitness; cardiometabolic risk; gut microbiota
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Metabolic Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be drawn by venous puncture for the measurement of different blood parameters (routine biochemistry, glycosylated hemoglobin, hemogram, hormones and exosomes). A clinical staff will take blood samples from a forearm vein after 8-10 hours of fasting. The sample will be collected in three Vacutainer plasma separator tubes anticoagulated with EDTA or heparin (5ml per tube) and one Vacutainer serum separator tube (10ml). Blood samples will be centrifuged for separation of plasma and serum, which will be stored at -80 °C until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- HIIT+Diet: High-Intensity Interval Training (HIIT) and Nutritional education
  Interventions: Other: No intervention
- MICT+Diet: Moderate-Intensity Continuous Training (MICT) and Nutritional education
  Interventions: Other: No intervention
- HIIT+NoDiet: High-Intensity Interval Training (HIIT) without Nutritional education. The HIIT training consisted of 3 sessions per week in a cycle ergometer, with 1-2 days off between sessions, during a total of 12 weeks under the supervision of a personal trainer. HIIT program consisted of 10 series of 1 min duration at 90% of peak power output, with 60 seconds of rest between sets (estimated total time of the session: 25 minutes).
  Interventions: Other: No intervention
- MICT+NoDiet: Moderate-Intensity Continuous Training (MICT) without Nutritional education. The MICT training consisted of 3 sessions per week in a cycle ergometer during 50 min at moderate intensity, with 1-2 days off between sessions, during a total of 12 weeks under the supervision of a personal trainer.
  Interventions: Other: No intervention
- Diet+NoExercise: Nutritional education without Exercise. The education intervention consisted of individual nutritional counselling. The nutritional education program was conducted every 2 weeks for 12 consecutive weeks, with 20-min counselling sessions by an experienced nutritionist. Participants were provided with an introduction (in an easy-to-understand manner) regarding the association between T2DM, gut microbiome and dietary habits. Firstly, the diet of the patient should be analysed, to determine which aspects can be improved, such as, total calories intake, amount and types of carbohydrates (highlighting the relevance of fibre), etc. Moreover, some suggestions about the combination of foods and culinary technical in order to manage the glycaemic index of foods were provided.
  Interventions: Other: No intervention
- Control group: Neither exercise nor nutritional education
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The study sample is divided into the six intervention groups of the EDUGUTION study (ClinicalTrials.gov Identifier: NCT05261373), although participants do not receive intervention in the present study, as only a description of the sample is made one year after the EDUGUTION study from a longitudinal perspective.

SUMMARY:
This longitudinal design study is a continuation of the EDUGUTION project (Ref: PID2019-110063RA-I00; Clinical Trial: NCT05261373), a randomized controlled trial that was approved by the Clinical Research Ethics Committee of Cadiz (Registration No. 92.21; PEIBA No. 1026-N-21) in 2021. The aim of this study was to determine the benefits of three months of intervention with physical exercise and nutritional counseling on health in patients with type 2 diabetes.

Specifically, the aim of the present longitudinal study is to analyze the possible changes that may have occurred in the health and lifestyle habits of the subjects of the EDUGUTION project one year after the end of the study. The tests to be performed are the following: 1) Analysis of sociodemographic information, diet and habits and quality of life with previously validated questionnaires, 2) Fasting blood collection, 3) Anthropometric and body composition assessment, 4) Assessment of physical fitness: manual grip strength and maximal oxygen uptake test.

On the same day in the morning, participants will have to go to the University Hospital of Puerto Real and to the Exercise Physiology Laboratory of the Faculty of Education Sciences of the Puerto Real Campus of the University of Cadiz, one year after the end of the EDUGUTION study. Since there is no intervention, the duration of the study is a single day. In this study 120 patients will participate, the same patients who were included based on the inclusion and exclusion criteria and who completed the EDUGUTION study intervention one year earlier.

DETAILED DESCRIPTION:
1. Sociodemographic Information and Questionnaires

   Sociodemographic information will include gender, age, ethnicity, education, employment and position in the organizational hierarchy, household composition (and person responsible for food shopping and cooking), marital status and information on urban or rural place of residence. With respect to the questionnaires, the following will be included:

   I) Adherence to the Mediterranean diet: the Mediterranean dietary pattern will be determined by a trained professional in a face-to-face interview. It will be established by means of a brief 14-item tool validated in Spanish population. Each question has a score of 0 or 1, since the values of the questionnaire range from 0 to 14. The higher the score, the greater the adherence to the Mediterranean dietary pattern.

   II) Quality of life: Self-reported quality of life will be recorded by applying the Short Form 36-health survey (SF-36) questionnaire previously validated in Spain. The SF-36 is a generic measure of quality of life and has been evaluated for a wide variety of medical conditions, including diabetes. The SF-36 includes 36 questions assessing 8 subscales, scores for each scale range from 0 to 100, with higher scores indicating a higher level of function or well-being.

   III) Bristol Scale: The Bristol visual stool chart will be used to classify stool form and condition, which classifies human stool form into seven groups, with 0 being the major constipation group and 7 being the major diarrhea group.

   IV) Sleep quality: The Pittsburgh sleep quality index previously validated in Spain will be used. The r-MEQ (reduced Morningness-Eveningness Questionnaire) of circadian rhythms will also be used.
2. Blood collection

   Participants will go to the University Hospital of Puerto Real coordinated by Dr. Florentino Carral in a fasting situation for the extraction of blood by venous blood for the measure of different blood parameters (biochemical parameters, glycosylated hemoglobin, hormones and exosomes). A clinical staff will take blood samples from a forearm vein after 8-10 hours of fasting. The sample will be collected in three Vacutainer plasma separator tubes anticoagulated with EDTA or heparin (5ml per tube) and one Vacutainer serum separator tube (10ml). Blood samples will be centrifuged for separation of plasma and serum, which will be stored at -80 °C until analysis. Plasma glucose and insulin concentrations will be determined by ELISA. These measurements will be used to calculate the HOMA-IR (Homeostatic Model Assessment for Insulin Resistance).
3. Anthropometry and body composition

   Subsequently, participants will have to go to the exercise physiology laboratory at the UCA in Puerto Real on an empty stomach. First, anthropometry measurements (height and body circumferences) and body composition (weight, body fat, muscle mass and body fluids) will be taken using previously validated 8-electrode multifrequency bioimpedance (TANITA- MC780MA). Patients will wear short, light clothing and assume a specific posture according to the manufacturer's instructions. In addition, 24 hours before the measurement, the following considerations will be followed: (i) refrain from physical exercise, (ii) do not drink alcoholic beverages, (iii) do not drink energy drinks and (iv) fast for at least 8 hours. Participants should urinate just before the measurement to ensure the elimination of body fluids.
4. Physical fitness: Muscle strength and cardiorespiratory fitness.

Finally, two physical fitness measurements will be performed in the same laboratory. First, muscle strength will be assessed by a manual grip test with a TKK-5401 digital hand-held dynamometer. Cardiorespiratory fitness will be assessed by an incremental test to exhaustion on a cycloergometer using a Jaeger MasterScreen CPX® gas analyzer (CareFusion, San Diego, USA). The test will start with a load of 30W in women and 50W in men, increasing 20W every minute until reaching maximal exhaustion to know the VO2max (maximal oxygen uptake). A pedaling cadence of over 70 rpm should be maintained throughout the test. During the stress test, Dr. Jose Maria Martin Cano (collegiate number: 111108959) will control the heart rate and vital signs to prevent any risk in the test or if there is any emergency situation.

At the end of the measurements, a detailed report with the results of the study will be given to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Non smoking
* Non-alcoholic (<3 standard drinks per day)
* Body mass index >25 kg/m maintaining the habitual dietary patterns without a body mass reduction higher than 2% during the last 6 months
* Not being insulin dependent
* Absence of injury, disease or disability or other known medical condition which could affect the ability to successfully participate in physical exercise tests
* Absence of cardiovascular disease (angina, peripheral or cerebro-vascular disease).
* Absence of neurologic and psychiatric diseases.
* Absence of respiratory diseases (pulmonary hypertension, Chronic obstructive pulmonary disease, etc.).
* Absence of other metabolic diseases (hyper/hypo parathyroidism, hyper/hypothyroidism, Cushing's disease, Type 1 diabetes, etc.)
* Absence of active inflammatory bowel disease
* Absence of kidney disease
* Absence of tumours
* Absence of coagulation dysfunction
* Not under treatment with medications k known to affect glucose metabolism, recent steroid treatment (within 6 months), or hormone replacement therapy
* Be able to understand a communication in Spanish or English.

Exclusion Criteria:

* Failure to complete the EDUGUTION study measurements and the intervention.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The sample of the present study consisted of adults (40-55 years) with type 2 diabetes mellitus or pre-diabetes. Patients must not be insulin dependent and all must be overweight/obese and sedentary people.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessed changes in Plasma Insulin | 1 year
  The ELISA technique will be used to determine the concentration of plasma insulin (mU/L) in a fasting situation.
Assessed changes in Plasma Glucose | 1 year
  Plasma glucose (mg/dL) will be analysed in a fasting situation.
Assessed changes in Glycosylated haemoglobin | 1 year
  Glycosylated haemoglobin (%) will be analysed in a fasting situation with the ADAMS™ A1C HA-8180V.
Assessed changes in Insulin Resistance | 1 year
  The Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) will be calculated using the glucose and insulin variables (HOMA-IR = fasting glucose (mg/dL) x fasting insulin (mU/L)/405).
Assessed changes from Body composition: Fatmass and Fat-free mass | 1 year
  Body composition will be estimated using a multifrequency bioimpedance of 8 electrodes previously validated (TANITAMC780MA). The calculation of impedance can estimate the fat mass and fat-free mass in kilograms. The patients will wear light clothing and will assume a posture in accordance with the manufacturers' instructions. Other previous considerations will be followed 24 hours before the measure: (i) to refrain from vigorous exercise, (ii) to take alcoholic drinks, (iii) to take energy drinks, and (iv) to be in a fasting state for at least 8 hours.
Assessed changes in Muscle Strength | 1 year
  Muscle strength will be assessed by a manual grip test with a TKK-5401 digital hand-held dynamometer.
Assessed changes from cardiorespiratory fitness | 1 year
  Cardiorespiratory fitness will be assessed by an incremental test to exhaustion on a cycloergometer using a Jaeger MasterScreen CPX® gas analyzer (CareFusion, San Diego, USA). The test will start with a load of 30W in women and 50W in men, increasing 20W every minute until reaching maximal exhaustion to know the VO2max (maximal oxygen uptake). A pedaling cadence of over 70 rpm should be maintained throughout the test. During the stress test, Dr. Jose Maria Martin Cano (collegiate number: 111108959) will control the heart rate and vital signs to prevent any risk in the test or if there is any emergency situation.

SECONDARY OUTCOMES:
Assessed changes from Sociodemographic situation | 1 year
  Sociodemographic information will include gender, age, ethnicity, education, employment and position in the organizational hierarchy, household composition (and person responsible for food shopping and cooking), marital status and information on urban or rural place of residence.
Assessed changes from self-reported quality of life | 1 year
  Self-reported quality of life will be registered by applying the Short Form 36-health survey (SF-36) questionnaire previously validated in Spain. The SF-36 is a generic measure of quality of life and has been evaluated for a wide variety of medical conditions, including diabetes. The SF-36 includes 36 questions that evaluate 8 subscales, scores for each scale range from 0 to 100, with higher scores indicating higher level of function or wellbeing. The physical component summary is derived from the 4 subscales of physical functioning, role physical, bodily pain, and general health; while the mental component summary is derived from the subscales of vitality, social functioning, role emotional, and mental health.
Assessed changes from Mediterranean diet adherence | 1 year
  The Mediterranean dietary pattern will be determined by a trained professional in a face-to-face interview. It will be established by means of a brief 14-item tool validated in Spanish population. Each question has a score of 0 or 1, since the values of the questionnaire range from 0 to 14. The higher the score, the greater the adherence to the Mediterranean dietary pattern.
Assessed changes in Stool status | 1 year
  The Bristol visual stool chart will be used to classify stool form and condition, which classifies human stool form into seven groups, with 0 being the major constipation group and 7 being the major diarrhea group.
Assessed changes in Sleep quality | 1 year
  The Pittsburgh Sleep Quality Index (PSQI) previously validated in Spain will be used. The measure consists of 19 individual items, creating 7 components that produce one global score.
Assessed changes in Circadian Rhythms | 1 year
  The r-MEQ (reduced Morningness-Eveningness Questionnaire) of circadian rhythms will be used. Total scores of the 5-item rMEQ range from 4 to 26, whereby a higher score indicates a morningness.